CLINICAL TRIAL: NCT06165653
Title: An Interventional Trial Using Guided Meditation During Radiation Therapy for Brain Tumors
Brief Title: Guided Meditation During Radiation Therapy for Brain Tumors
Acronym: Med-RT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI167297
Record Dates: First submitted 2023-11-10; First posted 2023-12-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Meditation Intervention (Experimental)
  Interventions: Behavioral: 5-Minute, Audio-Recorded Guided Mediation Practice
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: 5-Minute, Audio-Recorded Guided Mediation Practice — Five different meditation practices will be provided, all of which have been validated in prior research.
  * The Body Scan practice consists of instruction in how to direct non-judgmental attention to different regions of the body
  * The Mindful Breathing practice consists of focused attention on the breath and metacognitive monitoring and acceptance of discursive thoughts, negative emotions, and body sensations
  * The Mindfulness of Discomfort practice consists of instruction in how to "zoom in" to deconstruct discomfort and map each feelings' spatial location, use mindful breathing to "zoom out" and broaden the field of awareness to include neglected sensory elements, and shift attention from unpleasant feelings to neutral/pleasant sensations or experiences
  * The Savoring practice consists of instruction in identifying and amplifying pleasant memories
  * The Loving-Kindness practice consists of instruction in cultivating feeling of warmth and compassion toward the self and others
  Arms: Guided Meditation Intervention

SUMMARY:
The goal of this interventional treatment study is to assess the anxiolytic effect of providing guided meditation during radiation treatment (RT) in patients with brain tumors.

The main question it aims to answer is:

• What is the change in acute anxiety in participants receiving the mindfulness intervention during radiation therapy compared to standard of care control conditions?

Participants will be asked to participate in a 5-minute, audio-recorded mindfulness practice that will be played during the administration of each RT session. Researchers will compare this intervention to standard of care (no intervention) during RT.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years.
* Radiologically confirmed tumor of the brain. Note: Participants may have tumor resected after diagnosis.
* Eligible to undergo radiation treatment for brain tumor for 25-33 treatments.
* Willing to participate in either the guided meditation or standard of care control arm, regardless of treatment assignment.
* Karnofsky performance score ≥ 60 or ECOG performance score ≤ 2.
* MoCA mini score ≥ 11
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Active suicidal ideation or active psychotic state in the opinion of the investigator.
* An unstable illness that, in the opinion of the investigator, would interfere with study treatment.
* Prior radiation therapy to the brain.
* Inability to understand and/or speak the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in acute anxiety, measured by score on individual item derived from GAD-2, in participants receiving mindfulness intervention during RT compared to standard of care control conditions. | 7 weeks
  To assess the acute anxiolytic effects of a brief mindfulness intervention during RT for brain tumor patients with mask anxiety.
  Acute anxiety during RT will be measured each RT visit with an individual item ("How nervous, anxious or on edge do you feel right now?" scored on a 0-10 scale) derived from the Generalized Anxiety Disorder 2-item (GAD-2) scale, "0" meaning "Not at All" and "10" meaning "Very Much") measured before and after RT. The change from before to after RT will be averaged over all RT visits.

SECONDARY OUTCOMES:
Change in anxiety in everyday life in participants receiving mindfulness intervention during RT compared to standard of care, measured using the total score of the GAD-2 scale prior to RT | 7 weeks
  To assess the distal anxiolytic effects of a brief mindfulness intervention during RT for brain tumor patients with mask anxiety.
  Anxiety in everyday life will be measured using the total score of the Generalized Anxiety Disorder 2-item (GAD-2) scale prior to RT (minumum value 0, maximum value 6, score of 3 or higher considered clinical.) This will be measured once a week during RT.
Change in anxiety during RT and in everyday life as measured by the modified MPoD | 7 weeks
  To determine whether the brief mindfulness intervention during RT increases brain tumor patients' state mindfulness and whether the degree of changes in state mindfulness during RT predict decreases in acute anxiety and anxiety in daily life.
  Modified Metacognitive Processes of Decentering Scale (MPoD) consists of 4 items scored on a 0-10 scale, "0" meaning "Not at All" and "10" meaning "Very Much".
Change in self transcendence and the magnitude/degree of change in self transcendence as measured by total score of the Nondual Awareness Dimensional Assessment (NADA.) | 7 weeks
  To determine whether the brief mindfulness intervention during RT increases brain tumor patients' self transcendence and whether the degree of changes in self transcendence during RT predict decreases in anxiety in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burt, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No